CLINICAL TRIAL: NCT03912103
Title: An Interdisciplinary Deprescribing and Medication Optimization Intervention in an Integrated Outpatient Department: a Randomized Controlled Pilot Trial (FMA-CPH)
Brief Title: Interdisciplinary Medication Review Interventions in an Integrated Outpatient Department.
Acronym: FMA-CPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Hovedstadens Apotek (Other Government)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Anissa Aharaz, Clinical pharmacist, Region Hovedstadens Apotek
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VD-2019-09
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2019-03

CONDITIONS: Comorbidity; Multimorbidity; Drug Prescribing; Cognitive Impairment; Language Problems
Keywords: Deprescibing; Multimorbidity/comorbidity; Knowledge; Interdiciplinary intervention; Medication information; Motivation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Interdisciplinary medicine intervention focused on deprescribing and medication optimization. The control group receives standard care.
  Finally we investigate the number of patients who have completed at least one deprescribing and/or medication optimization in each group.
Who Masked: Outcomes Assessor
Masking Description: The evaluation of completed deprescribing and/or medication optimization are performed by two blinded assessors (senior clinical pharmacist and/or medical physicians).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdiciplinary medication review intervention (Active Comparator): The clinical pharmacist perform medication review and presents medication interventions orally and written to the physician. The physician perform the changes and inform the patient about the changes. 7 days after intervention the patient receives a follow up phone call from the pharmacist about the medication interventions. If the pharmacist during the follow up phone call identify any complications due to compliance/add on/deprescribing the pharmacist uses motivational conversation to come to a solution.14 days after the beginning of the intervention the patients knowledge about their medication and satisfaction with medication information is investigated by a phone questionnaire and measured on a Likert scale (1-5). 30 days after the beginning of the intervention the pharmacist collect an updated medication history. Finally we investigate the number of patients who have completed at least one deprescribing and/or medication optimization in each group.
  Interventions: Other: Interdisciplinary Deprescribing and Medication Optimization Intervention
- Control group (No Intervention): Standard treatment without a medication review and follow up related to medication changes (standard treatment).14 days after the enrollment the patients knowledge about their medication and satisfaction with medication information is investigated by a phone questionnaire measured on a Likert scale (1-5). 30 days after the enrollment the pharmacist collect an updated medication history.Finally we investigate the number of patients who have completed at least one deprescribing and/or medication optimization in each group

INTERVENTIONS:
Other: Interdisciplinary Deprescribing and Medication Optimization Intervention — as current
  Arms: Interdiciplinary medication review intervention

SUMMARY:
Inappropriate medication prescribing is highly prevalent among comorbid medical patients and leading to adverse drug events (ADE), re-admissions, quality of life and mortality. Thus, the aim of this study is primary to investigate the feasibility of a interdisciplinary intervention focused on deprescribing and medication optimization in the Integrated Outpatient Department at Copenhagen University Hospital, Amager, Denmark.

Participants in the intervention group receives a medication review by a clinical pharmacist and physician with a follow up after 7 and 30 days. The control group receives standard care.

DETAILED DESCRIPTION:
The FMA-CPH trial is designed as a single-blinded randomized controlled pilot trial starting at the first consultation and end 30 days after.

Patients that meet all inclusion criteria and none of the exclusion criteria are invited to participate. After signing a written informed consent, the participants are block randomized to either the intervention or control group.

Medication prescription for comorbid patients is challenging and may be attributed to marked inter-individual variations in general health, organ function, pharmacokinetic and pharmacodynamic properties, biological age and physical performance. The intervention group receive a medication review.

It is hypothesized that the intervention is feasible and more patients in the intervention group will complete ≥1 deprescribing and/or ≥1 medication optimization 30 days after the beginning of the intervention than the patients in the control group.

Secondary it is hypothesized the patients in the intervention group:

A. Complete more deprescribing compared to the control group (30 days after intervention) B. Complete more medication optimization compared to the control group (30 days after intervention) C. Have a higher knowledge about own medication (14 days after intervention) D. Have a higher level of satisfaction with medication information (14 days after intervention)

ELIGIBILITY:
Inclusion Criteria:

* Consultation at Integrated Outpatient Department subacute track
* Multi morbidity/Comorbidity
* Drug Prescribing
* Mentally fresh
* Understand and speak Danish

Exclusion Criteria:

* Unable to cooperate cognitively
* Language problems
* Admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of a deprescribing and medication optimization: Number of patients who complete ≥1 deprescribing and/or ≥1 medication optimization 30 days after enrolment in each group. | Baseline to 30 days after enrolment
  Number og patients who complete ≥1 deprescribing and/or ≥1 medication optimization 30 days after enrolment in the study.

SECONDARY OUTCOMES:
Difference in patients between the two groups who completed ≥1 deprescribing and/or dose reduction 30 days after enrolment. Difference as %. | Baseline to 30 days after enrolment
  Number of patients in the intervention group who complete ≥1 deprescribing and/or dose reduction than control group 30 days after enrolment in each group. Difference expressed as a percentage.
Difference in patients between the two groups who completed ≥1 medication optimization 30 days after enrolment in each group. Difference as % | Baseline to 30 days after enrolment
  Number of patients in the intervention group who complete ≥1 medication optimization more than control group 30 days after enrolment in each group. Difference expressed as a percentage.
Difference in Knowledge between the two groups who gains more knowledge about their medication measured by ≥1 point on Likert scale (1-5 p). | Baseline to 14 days after enrolment
  Number of patients in the intervention group who gains more knowledge about their medication measured by ≥1 point more than patients in the control group measured in difference in points on Likert scale (1-5 points). Where 5 points indicates high knowledge and 1 point is no knowledge. Difference expressed as a percentage
Difference in patients who are satisfied with medication information measured by ≥1 point on Likert scale (1-5 p). | Baseline to 14 days after enrolment
  Number of patients in the intervention group who are more satisfied with medication information given by the Interdisciplinary team measured by ≥1 point than patients in control group measured in difference in points on Likert scale (1-5p). Where 5 points indicates high knowledge and 1 point is no knowledge. Difference expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Helle Ø McNulty, cand pharm, Study Director — Region Hovedstadens Apotek; Charlotte Treldal, Phd, Study Chair — Region Hovedstadens Apotek
Locations (1):
- Capital Regional Hospital, Amager, Integrated Outpatient Department, Copenhagen, Denmark